CLINICAL TRIAL: NCT06369805
Title: EVALUATION DE L'AIDE AU DIAGNOSTIC PAR BIOMARQUEURS SANGINS CHEZ DES PATIENTS SOUFFRANT DE DEPRESSION SUIVIS EN AMBULATOIRE
Brief Title: EVALUATION OF BLOOD BIOMARKER-BASED DIAGNOSTIC AID IN OUTPATIENTS SUFFERING FROM DEPRESSION
Status: Completed | Type: Observational
Sponsor: Les Toises - Psychiatry and Psychotherapy Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00731
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder; Bipolar Disorder; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- one group
  Interventions: Other: there is no intervention

INTERVENTIONS:
Other: there is no intervention — there is no intervention

SUMMARY:
This is an observational (non-interventional) study, carried out in an outpatient setting, which involves a blood sampling. The primary objective of this study is to confirm the association between the EDIT-B® editing signature and early unipolar or bipolar differentiation. Results of this research may provide an aid to early diagnosis and guide clinical practice towards individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

Adult outpatients suffering from depression and/or bipolar disorders who gave their written informed consent to participate in the present study

Exclusion Criteria:

Any patient without capacity of discernment or with harmful use of psychoactive substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients suffering from depression and/or bipolar disorders
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Psychiatric symptomatology | Once
  self- and hetero-psychiatric scales

CONTACTS AND LOCATIONS:
Locations (1):
- Les Toises - Psychiatry and Psychotherapy Center, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No